CLINICAL TRIAL: NCT05039879
Title: Life Improving Factors After a Hip Fracture
Acronym: LIFF
Status: Completed | Type: Observational
Sponsor: Wageningen University (Other)
Collaborators: Rijnstate Hospital (Other)
Responsible Party: Principal Investigator, Hugo Wijnen, Drs., Rijnstate Hospital
Other Study IDs: 2021-1814
Record Dates: First submitted 2021-07-21; First posted 2021-09-10 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Hip Fractures; Older Adults
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary objective of the proposed research is to investigate the association between protein intake and nutritional status with bone health and physical functioning in older hip fracture patients. In addition, it will be investigated which patient characteristics and modifiable factors can predict mobility, clinical frailty, living situation and mortality. This study will be a 3-month prospective cohort study in adults aged 70 years and older with an acute hip fracture. This study will lead to knowledge about how protein intake and nutritional status in combination with patient characteristics can predict the degree of recovery (bone health and physical functioning) 3 months after the hip fracture. Knowledge on factors related to recovery can contribute to an improved and shorter rehabilitation in the future, which results in a reduction of health care costs.

DETAILED DESCRIPTION:
Only half of the patients with an acute hip fracture regain their pre-fracture functional level and 24% dies within the following year. Identifying and targeting modifiable risk factors for optimal recovery after a hip fracture is therefore essential. These factors include protein intake and nutritional status, which may affect markers of bone health and physical functioning and thereby influence recovery.

Measurements will be performed at baseline (within 5 days after the hip surgery) and after 3 months during an outpatient clinic visit for the evaluation of the hip fracture surgery. A total of 95 older adults (aged 70 years or older) recovering from an acute hip fracture will be recruited from Rijnstate hospital.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 70 years
* Community-dwelling
* Proximal femur fracture: femoral neck fracture/ pertrochanteric fracture, subtrochanteric fracture
* Able to give informed consent
* Pre-fracture Clinical Frailty Scale 3-6

Exclusion Criteria:

* Pathological fracture or periprosthetic fracture
* Current participation in scientific research that interferes with the proposed study
* History of dementia
* No permission to request information from the general practitioner/ treating specialist(s) about medical history, medication use, liver and kidney values, and details about the broken hip

Min Age: 70 Years | Sex: All
Age Groups: Older Adult
Study Population: Older adults aged 70 years or older recovering from an acute hip fracture
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2021-09-06 (Actual); Primary Completion 2022-11-29 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Protein intake | Baseline
  Dietary protein intake will be recorded using a protein screener which gives an indication of protein intake in g/d. Based on the past 4 weeks.
Protein intake | Three months
  Dietary protein intake will be recorded using a protein screener which gives an indication of protein intake in g/d. Based on the past 4 weeks.
Nutritional status | Baseline
  Using the Mini Nutritional Assessment Short Form. Subjects will be classified as having a normal nutritional status (12-14 points), having a risk of malnutrition (8-11 points), or being undernourished (0-7 points).
Nutritional status | Three months
  Using the Mini Nutritional Assessment Short Form. Subjects will be classified as having a normal nutritional status (12-14 points), having a risk of malnutrition (8-11 points), or being undernourished (0-7 points).
Procollagen type 1 N propeptide | Baseline
  Bone turnover marker, in serum
Procollagen type 1 N propeptide | Three months
  Bone turnover marker, in serum
C-terminal telopeptide of type I collagen | Baseline
  Bone turnover marker
C-terminal telopeptide of type I collagen | Three months
  Bone turnover marker
Calcaneus quantitative ultrasound parameters | Baseline
  Ultrasound of the calcaneus which gives an indication of the bone density. Device yields the following two parameters: speed of sound (SOS) and broadband ultrasound attenuation (BUA), which can be combined to get the Stiffness Index (SI).
Calcaneus quantitative ultrasound parameters | Three months
  Ultrasound of the calcaneus which gives an indication of the bone density. Device yields the following two parameters: speed of sound (SOS) and broadband ultrasound attenuation (BUA), which can be combined to get the Stiffness Index (SI).
Insulin-like growth factor 1 | Baseline
  In serum
Insulin-like growth factor 1 | Three months
  In serum
Parathyroid hormone levels | Baseline
  In serum
Parathyroid hormone levels | Three months
  In serum
Handgrip strength | Baseline
  Using the Martin vigorimeter
Handgrip strength | Three months
  Using the Martin vigorimeter
Grip work | Baseline
  Using the Martin vigorimeter
Grip work | Three months
  Using the Martin vigorimeter

SECONDARY OUTCOMES:
Appendicular skeletal muscle mass | Baseline
  Using bioimpedance spectroscopy
Appendicular skeletal muscle mass | Three months
  Using bioimpedance spectroscopy
Mobility | Baseline
  Pre-fracture mobility will be assessed with the pre-fracture mobility scale (PMS). The PMS classifies the patient as independent walker, walk with rollator, in a wheelchair or bedridden.
Mobility | Three months
  Mobility at 3 months will be assessed with the Functional Ambulation Categories (FAC). The FAC is scaled from 0 to 5, in which zero means that patient cannot walk or need at least two persons to help and five means independent walker.
Frailty | Baseline
  Frailty will be assessed with the Clinical Frailty Scale. This scale is graded from 1 to 9 in which level 1 represents 'very fit' and level 9 'terminally ill'.
Frailty | Three months
  Frailty will be assessed with the Clinical Frailty Scale. This scale is graded from 1 to 9 in which level 1 represents 'very fit' and level 9 'terminally ill'.
Bodyweight | Baseline
  Bodyweight (kg) will be measured with a calibrated sitting weighing scale.
Bodyweight | Three months
  Bodyweight (kg) will be measured with a calibrated sitting weighing scale.
Barthel Index | Baseline
  This questionnaire determines the degree of (physical or verbal) help a person needs to perform general daily activities. It is graded from 0 (person is completely dependent on others) to 20 (person is completely independent).
Barthel Index | Three months
  This questionnaire determines the degree of (physical or verbal) help a person needs to perform general daily activities. It is graded from 0 (person is completely dependent on others) to 20 (person is completely independent).

CONTACTS AND LOCATIONS:
Overall Officials: Hugo Wijnen, Principal Investigator — Hospital Rijnstate
Locations (1):
- Rijnstate Hospital, Arnhem, Netherlands

IPD SHARING:
Plan to Share IPD: No